CLINICAL TRIAL: NCT05124886
Title: Gut Kidney Axis in Enteric Hyperoxaluria: A Clinical Prospective Study of the Effects of the Microbiome on Urinary Oxalate in Participants With Enteric Hyperoxaluria Fed a Moderate Oxalate Diet
Brief Title: Gut Kidney Axis in Enteric Hyperoxaluria
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-01274; R01DK128842 (NIH)
Record Dates: First submitted 2021-11-03; First posted 2021-11-18 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Enteric Hyperoxaluria
MeSH Terms: interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Controls (Active Comparator)
  Interventions: Other: Moderately High Oxalate (MOx) Diet
- Enteric Hyperoxaluria (Experimental)
  Interventions: Other: Moderately High Oxalate (MOx) Diet

INTERVENTIONS:
Other: Moderately High Oxalate (MOx) Diet — Diets will contain 16% protein, 30% fat, and 54% carbohydrate, and are controlled in the amounts of calcium (400mg), oxalate (250mg), ascorbic acid (50mg), fiber (30 grams) and, other nutrients. Each controlled diet will be consumed for four days. On days of controlled diets, subjects will be provided with 2 liters of bottled water per day to ensure adequate hydration. After the controlled diet period, there will be a three-day washout period, where participants will consume Ad-lib diets supplemented with a daily intake of oxalate in the form of cooked spinach to be taken with breakfast daily for a total of 2 weeks.

SUMMARY:
40 subjects with a confirmed diagnosis of IBD or >6 months post-RYGB with a diagnosed USD event or kidney stone on imaging within the past three years and 40 healthy controls will be administered a high oxalate diet on Days 0-3 and Days 21-24 with a washout period on Days 4-7 and will be administered 250mg sodium oxalate on Days 8-20, via prepared spinach, from Weil Cornell Medicine's Clinical and Translational Science Center. Subjects will partake in four stool collections, four 24-h urine collections, two blood collections, and four sets of colonic permeability testing.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Subjects > 18 years and < 80 years of age
* a confirmed diagnosis of IBD or > 6 months post- RYGB, with a diagnosis USD event (renal colic with spontaneous stone passage, emergency room visits, or urological interventions) or have kidney stone on imaging (CT, MRI, or US) in the previous three years.
* We will include all racial and ethnic groups, and both men and women.

In order to be eligible in this study as a healthy control, an individual must meet all of the following criteria:

* Subjects > 18 years and < 80 years of age
* Healthy controls with no chronic diseases, not on any chronic medications, no history of GI pathology, or urinary stone disease (USD).
* We will include all racial and ethnic groups, and both men and women.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* pregnant or nursing women and people with any medical, psychiatric, debilitating disease/disorder or social condition that, in the judgment of the investigator, would interfere with or serve as a contraindication to adherence to the study protocol, ability to give ICF or complete the protocol.
* subjects with total and partial colectomy.
* subjects who received oral, intramuscular, or intravenous antibiotics within three months before screening.
* Patients with perianal disease usually receive recurrent antibiotics and, therefore, will be excluded from the study.
* patients with an ongoing symptomatic IBD flare or a flare within the previous three months
* patients with estimated glomerular filtration rates (eGFR) < 60 ml/min/1.73 m2 calculated by the CKD-EPI equation measured anytime within the preceding year.

An individual who meets any of the following criteria will be excluded from participation in this study as a healthy control:

* pregnant or nursing women and people with any medical, psychiatric, debilitating disease/disorder or social condition that, in the judgment of the investigator, would interfere with or serve as a contraindication to adherence to the study protocol, ability to give ICF or complete the protocol.
* subjects with total and partial colectomy.
* subjects who received oral, intramuscular, or intravenous antibiotics within three months before screening.
* Patients with perianal disease usually receive recurrent antibiotics and, therefore, will be excluded from the study.
* patients with an ongoing symptomatic IBD flare or a flare within the previous three months
* patients with estimated glomerular filtration rates (eGFR) < 60 ml/min/1.73 m2 calculated by the CKD-EPI equation measured anytime within the preceding year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Urinary Oxalate Levels (UOx) | Day 2-3
  UOx will be quantified in 24-h samples
Urinary Oxalate Levels (UOx) | Day 23-24
  UOx will be quantified in 24-h samples

SECONDARY OUTCOMES:
Total Fecal Oxalate Levels | Day 2-3
Total Fecal Oxalate Levels | Day 14
Total Fecal Oxalate Levels | Day 23-24
Urinary Calcium Levels | Day 2-3
Urinary Calcium Levels | Day 23-24
Sucralose Levels | Day 2-3
Sucralose Levels | Day 23-24
Calcium Oxalate (CaOx) Supersaturation Levels | Day 2-3
Calcium Oxalate (CaOx) Supersaturation Levels | Day 23-24
Plasma Oxalate Levels | Day 2-3
Plasma Oxalate Levels | Day 23-24

CONTACTS AND LOCATIONS:
Overall Officials: Lama Nazzal, MD, Study Chair — NYU Langone Health; David Goldfarb, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected for this study will be analyzed and stored at the Nazzal-hyperoxaluria data repository. After the study is completed, the de-identified, archived data will and stored at the Nazzal- hyperoxaluria data repository, under the supervision of Dr. Lama Nazzal, for use by other researchers including those outside of the study. Permission to transmit data to the Nazzal-hyperoxaluria data repository will be included in the informed consent.
  Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to lama.nazzal@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.